CLINICAL TRIAL: NCT07359404
Title: A Phase II Clinical Study of Sacituzumab Govitecan Combined With Bevacizumab for the Treatment of Patients With Metastatic Triple-Negative Breast Cancer
Brief Title: Sacituzumab Govitecan Plus Bevacizumab in Metastatic TNBC
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: YING FAN (Other)
Responsible Party: Sponsor-Investigator, YING FAN, Principal Investigator, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-Gilead2024-PT-0284
Record Dates: First submitted 2025-12-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — sacituzumab govitecan; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sacituzumab Govitecan + Bevacizumab (Experimental)
  Interventions: Drug: Sacituzumab Govitecan (SG); Drug: Bevacizumab

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG) — Administered via intravenous infusion on Day 1 and Day 8 of each 21-day cycle. In the Safety Run-in phase, the starting dose is 10 mg/kg, with a potential de-escalation to 7.5 mg/kg based on Dose-Limiting Toxicity (DLT). In the Expansion phase, patients receive the determined recommended dose
Drug: Bevacizumab — Administered by intravenous infusion on the first day of each 21-day cycle. In the safety trial phase, the starting dose is 7.5 mg/kg and can be reduced to 5 mg/kg depending on dose-limiting toxicity (DLT). During the expansion phase, patients receive the determined recommended dose

SUMMARY:
This is a single-arm, multicenter, Phase II clinical study aiming to explore the efficacy and safety of Sacituzumab Govitecan combined with Bevacizumab as a second-line or later treatment for patients with metastatic triple-negative breast cancer (mTNBC). The study will be conducted in 6-8 centers in China.

The study is divided into two phases: a Safety Run-in Phase and a Dose Expansion Phase.

In the Safety Run-in Phase (3-12 patients), three dose levels are planned to determine the recommended dose. The starting dose (Level 1) is Sacituzumab Govitecan 10 mg/kg (Days 1, 8) plus Bevacizumab 7.5 mg/kg (Day 1) every 21 days. Based on the occurrence of Dose-Limiting Toxicities (DLT) in the first cycle, the Safety Monitoring Committee (SMC) will decide whether to continue the current dose or de-escalate to Level 2 (Sacituzumab Govitecan 10 mg/kg + Bevacizumab 5 mg/kg) or Level 3 (Sacituzumab Govitecan 7.5 mg/kg + Bevacizumab 5 mg/kg).

In the Dose Expansion Phase, 40-50 patients will be enrolled to receive the combination therapy at the recommended dose determined in the run-in phase. Efficacy will be evaluated every 2 cycles according to RECIST 1.1, and safety will be assessed continuously until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged > 18 years.
2. Pathologically confirmed recurrent or metastatic Triple-Negative Breast Cancer (TNBC).
3. ER and PR negativity is defined as < 10% expression in tumor cells. HER2 negativity is defined as IHC 0, 1+, or IHC 2+ with FISH negative. Must have received at least one prior systemic therapy in the metastatic setting.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Life expectancy of more than 3 months.
6. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
7. Adequate organ function.
8. Sufficient washout period before screening (3 weeks from last chemotherapy, 4 weeks from last targeted therapy)

Exclusion Criteria:

1. Prior treatment with Sacituzumab Govitecan or Bevacizumab.
2. Uncontrolled central nerve
3. Presence of other primary malignancies.
4. Severe infection, severe cardiac disease, autoimmune disease, or other conditions deemed unsuitable for anti-tumor therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From start of treatment until disease progression or death, assessed up to approximately 32 months (based on study completion date of Dec 2026)
Incidence and Severity of Adverse Events (Safety) | From start of treatment through 90 days after the last dose of study drug.

SECONDARY OUTCOMES:
Objective Response Rate | From start of treatment until disease progression or intolerance, assessed every 2 cycles, assessed up to approximately 32 months
Overall Survival | From start of treatment until death, assessed up to approximately 32 months
Disease Control Rate | From start of treatment until disease progression or intolerance, assessed up to approximately 32 months
Duration of Response | From date of first response until disease progression or death,assessed up to approximately 32 months
6-month Progression-Free Survival Rate | At 6 months after treatment initiation
6-month Overall Survival Rate | At 6 months after treatment initiation

OTHER OUTCOMES:
Trop-2 Expression Level | From baseline up to approximately 32 months
  Assessment of Trop-2 expression in tumor tissue using Immunohistochemistry (IHC). Results are reported as Histochemical Score (H-score, ranging from 0 to 300). This measure will be analyzed to explore the association with efficacy outcomes (PFS, ORR).
UGT1A1 Genotype Status | From baseline up to approximately 32 months
  Assessment of UGT1A1 gene polymorphisms (e.g., 1, 28 alleles) in blood or tissue samples using PCR or sequencing. Results are categorized by genotype (e.g., homozygous wild-type, heterozygous, homozygous mutant). This measure will be analyzed to explore the association with safety outcomes (adverse events).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No